CLINICAL TRIAL: NCT00965562
Title: A Double-blind, Parallel Comparison of Fluoxetine, Calcium and Placebo for the Treatment of Moderate to Severe Premenstrual Syndrome (PMS)
Brief Title: Comparison of Fluoxetine, Calcium and Placebo for the Treatment of Moderate to Severe Premenstrual Syndrome (PMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donaghue Medical Research Foundation (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Kimberly Yonkers, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0001011511; NCT00683605 (obsolete NCT alias)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-02

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual syndrome; PMS; calcium
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Fluoxetine; Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I (Active Comparator): Fluoxetine
  Interventions: Drug: Fluoxetine
- II (Active Comparator): Calcium
  Interventions: Drug: Calcium
- III (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine 20 mg per day for 4 menstrual cycles. For the fifth menstrual cycle, all women will receive calcium. Women on Fluoxetine will continue taking it in addition to 1200mg of calcium.
  Other Names: Prozac
  Arms: I
Drug: Calcium — 1200 mg of calcium to be taken for 5 menstrual cycles.
  Arms: II
Drug: Placebo — For 5 cycles, women will receive placebo. At the end of the fourth cycle, all women will receive 1200 mg of calcium in addition to the placebo medication.
  Arms: III

SUMMARY:
The purpose of this study is to compare the efficacy of calcium carbonate to fluoxetine in the treatment of moderate to severe PMS. Second, to compare each active agent to a placebo control. Third, to evaluate the efficacy of each treatment for specific symptom clusters (i.e. affective and somatic). Fourth, to determine whether the addition of calcium to on going fluoxetine treatment leads to additional therapeutic benefit.

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo controlled, parallel study that will randomize 60 women at the Yale site into treatment. Participants will be screened at various collaborating ob-gyn centers for possible PMS symptoms, and direct referrals from the community will also be accepted. Subject participation length is about 7 months with 6 scheduled study visits.

Methodology: After successfully completing the screening and qualification phase, participants will be randomized to treatment at Visit 1 for 5 cycles of double-blind treatment. Participants will be evaluated monthly during the randomization phase for adverse events, concurrent medication, and primary and secondary efficacy variables.

.

ELIGIBILITY:
Inclusion Criteria:

* Female outpatients between the ages of 18 and 48 who are:

  * Menstruating
  * Meet criteria for moderate to severe PMS
  * Report PMS symptoms for at least 9 our of the 12 months prior to screening; 4) *Are using an adequate method of birth control.

Exclusion Criteria:

* Any candidate who:

  * Fulfills MINI (DSM-IV) criteria for a serious AXIS 1 disorder
  * Fulfills DSM-IV criteria during the charting phase consistent with a diagnosis of psychotic disorder, bipolar disorder or major depressive disorder
  * Has a severe, co-existing condition that, in the investigator's opinion, renders the patient unsuitable for the study
  * Poses a significant risk of suicide
  * Takes ongoing medication that could treat PMS symptoms
  * Has a history of hypersensitivity or adverse reaction to fluoxetine or calcium
  * Is lactating, pregnant or is planning to become pregnant during the course of the study.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2000-09; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Yonkers, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred through on-site screening in private gynecological practices and community advertisements. Recruitment occurred between 2001-2005 in Providence, Rhode Island and between 2001-2009 in New Haven, Connecticut. Potential subjects provided consent for screening and assessment.
Groups:
- I: Fluoxetine: Fluoxetine : Fluoxetine 20 mg per day for 4 menstrual cycles.
- II: Calcium: Calcium : 1200 mg of calcium to be taken for 4 menstrual cycles.
- III: Placebo: Placebo : For 4 cycles, women will receive placebo.
Period: Overall Study
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Started | 16 | 17 | 16
Women With at Least 2 Follow up Visits | 13 (3 patients with no follow up visits: 1 out of contact, 2 patient requests) | 13 (4 patients with no follow up visits: 2 out of contact, 2 patient requests) | 13 (3 patients with no follow up visits: 3 out of contact)
Women Who Participated Full Follow up | 6 (7 patients discontinued intervention: 2 out of contact, 4 patient requests, 1 suspended by IRB) | 10 (3 patients discontinued intervention: 1 out of contact, 2 patient requests) | 11 (2 patients discontinued intervention: 2 patient requests)
Completed | 13 (Participants who completed at least 2 visits were analyzed.) | 13 (Participants who completed at least 2 visits were analyzed.) | 13 (Participants who completed at least 2 visits were analyzed.)
Not Completed | 3 | 4 | 3
Not completed — Lost to Follow-up | 1 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants with at least 2 follow up visits were included in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Customized [Number; unit: participants]
  25-29 years old | 1 | 1 | 2 | 4
  30-39 years old | 11 | 6 | 7 | 24
  40-45 years old | 1 | 6 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 13 | 39
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 8 | 10 | 10 | 28
  Black | 1 | 0 | 0 | 1
  Hispanic | 1 | 0 | 1 | 2
  Other/Mixed | 2 | 1 | 1 | 4
  Not collected | 1 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 13 | 39
Marital Status [Number; unit: participants]
  Married | 7 | 8 | 9 | 24
  Single/Divorced/Widowed | 5 | 5 | 4 | 14
  Not collected | 1 | 0 | 0 | 1
Number of pregnancies [Number; unit: participants]
  0 pregnancies | 6 | 3 | 5 | 14
  1 pregnancy | 3 | 1 | 0 | 4
  2+ pregnancies | 4 | 9 | 8 | 21
Years with PMS [Number; unit: participants] — PMS= premenstrual syndrome.
  participants
    <4 years | 6 | 2 | 6 | 14
    5-10 years | 3 | 6 | 1 | 10
    >10 years | 3 | 5 | 6 | 14
    Number of years not collected | 1 | 0 | 0 | 1
Ever spoken to a doctor about PMS [Number; unit: participants] — PMS= premenstrual syndrome. Only participants who indicated that they had spoken to a doctor about their PMS were included in this affirmative measure.
  participants | 4 | 5 | 6 | 15
OB-GYN asked about PMS [Number; unit: participants] — PMS= premenstrual syndrome. Only participants who indicated that their OB-GYN had asked about PMS were included in this affirmative measure.
  participants | 2 | 5 | 2 | 9
Thought about getting help for PMS [Number; unit: participants] — PMS= premenstrual syndrome. Only participants who indicated that they had thought about getting help for their PMS symptoms were included in this affirmative measure.
  participants | 7 | 7 | 6 | 20
Concurrent oral contraceptive use [Number; unit: participants] — Only participants who indicated that they were concurrently taking contraceptives were included in this affirmative measure.
  participants | 4 | 3 | 3 | 10
Baseline Symptom Scores [Mean (Standard Deviation); unit: units on a scale] — IDS= sum of responses to 28 of 30 possible items each scored 0 to 3 points (0=least severe 84= most severe); PMTS= total score 10 items, each with 4 points (0 is no symptom and 40 total = most severe); CGI-S= illness severity (1=normal 7=among most critically ill) . The IDS, PMTS, and CGI-S were scored on the basis of severity during the prior premenstrual phase. DRSP= 21 items each with scale (1=no symptom 6=extreme); The DRSP score was generated by subtracting average follicular phase severity from average luteal phase severity, and averaging these phase change means across symptoms.
  units on a scale
    Inventory of Depressive Symptomatology (IDS-C30) | 31.85 (9.14) | 30.92 (7.62) | 28.85 (9.97) | 30.54 (5.17)
    Premenstrual Tension Syndrome-Observer (PMTS-O) | 24.15 (5.40) | 21.58 (3.73) | 20.85 (6.62) | 22.19 (3.11)
    Daily Record of Severity of Problems (DRSP) | 2.16 (0.86) | 1.12 (0.38) | 1.29 (0.60) | 1.52 (0.37)
    Clinical Global Impression - Severity (CGI-S) | 4.92 (0.95) | 4.46 (1.27) | 4.15 (1.28) | 4.51 (0.68)

OUTCOME MEASURES:

1. Secondary Outcome: Proportion of Participants With DRSP LOCF Response to Treatment (50% Improvement)
Description: DRSP: Daily Record of Severity of Problems, which combines responses to 21 items each with scale: 1=no symptoms, 6=extreme. LOCF: the last observation carried forward.
Time Frame: over duration of treatment, 4 menstrual cycles averaging 4 months after baseline visit
Population: Response analysis includes all data from all subjects with the last observation carried forward to Visit 5.
Measure: Number; unit: proportion of participants
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 10 | 12 | 12
proportion of participants | 0.80 | 0.42 | 0.42
Statistical Analysis 1: Comparison: I: Fluoxetine vs II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.15, Chi-squared

2. Secondary Outcome: Proportion of Participants With IDS LOCF Response to Treatment (50% Improvement)
Description: IDS: Inventory of Depressive Symptomatology: measures depressive symptoms during the previous premenstrual phase with high internal consistency: sum of responses to 28 of 30 possible items each scored 0 to 3 points with total scoring (0=least severe, 84=most severe). LOCF: last observation carried forward.
Time Frame: over duration of treatment, 4 menstrual cycles averaging 4 months after baseline visit
Population: Response analysis includes all data from all subjects with the last observation carried forward to Visit 5.
Measure: Number; unit: proportion of participants
Groups:
- III: Placebo: Placebo : For 5 cycles, women will receive placebo.
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 13 | 13 | 13
proportion of participants | 0.77 | 0.31 | 0.31
Statistical Analysis 1: Comparison: I: Fluoxetine vs II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.05, Chi-squared

3. Secondary Outcome: Proportion of Participants With PMTS LOCF Response to Treatment (50% Improvement)
Description: PMTS: Premenstrual Tension Syndrome (Observer Rating) Scale: a clinician-administered retrospective scale developed for the study of PMS, a sum of responses to 10 items each with 4 points (0=no symptoms, 40=most severe). LOCF: last observation carried forward.
Time Frame: over duration of treatment, 4 menstrual cycles averaging 4 months after baseline visit
Population: Response analysis includes all data from all subjects with the last observation carried forward to Visit 5.
Measure: Number; unit: proportion of participants
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 13 | 12 | 13
proportion of participants | 0.62 | 0.33 | 0.16
Statistical Analysis 1: Comparison: I: Fluoxetine vs II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.06, Chi-squared

4. Secondary Outcome: Proportion of Participants With DRSP Visit-wise Response to Treatment (50% Improvement)
Description: Visit-wise response considers participants who remained in the study until Visit 5 and provided data for the visit. DRSP = Daily Record of Severity of Problems, which combines responses to 21 items each with scale: 1=no symptoms, 6=extreme.
Time Frame: over duration of treatment from baseline to visit 5, including 4 menstrual cycles averaging 4 months after baseline visit
Population: For fluoxetine, calcium and placebo groups, 8, 11 and 12 participants remained in the trial until Visit 5. However, Visit 5 DRSP calendars were missing for an additional 3 subjects in the fluoxetine group and for one subject in each of the calcium and placebo cells.
Measure: Number; unit: proportion of participants
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 5 | 8 | 6
proportion of participants | 1.00 | 0.50 | 0.33
Statistical Analysis 1: Comparison: I: Fluoxetine vs II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.09, Chi-squared

5. Secondary Outcome: Proportion of Patients With IDS Visit-wise Response to Treatment (50% Improvement)
Description: Visit-wise response considers participants who remained in the study until Visit 5 and provided data for the visit.
  IDS = Inventory of Depressive Symptomatology: measures depressive symptoms during the previous premenstrual phase with high internal consistency, sum of responses to 28 of 30 possible items each scored 0 to 3 points with total scoring (0=no symptoms, 84=most severe).
Time Frame: as for outcome 4
Population: For fluoxetine, calcium and placebo groups, 8, 11 and 12 participants remained in the trial until Visit 5.
Measure: Number; unit: proportion of participants
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 8 | 11 | 12
proportion of participants | 1.00 | 0.36 | 0.33
Statistical Analysis 1: Comparison: I: Fluoxetine vs II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.005, Chi-squared

6. Secondary Outcome: Proportion of Patients With PMTS Visit-wise Response to Treatment (50% Improvement)
Description: Visit-wise response considers participants who remained in the study until Visit 5 and provided data for the visit. PMTS = Premenstrual Tension Syndrome (Observer Rating) Scale: a clinician-administered retrospective scale developed for the study of PMS, a sum of responses to 10 items each with 4 points (0=no symptoms, 40=most severe).
Time Frame: as for outcome 4
Population: For fluoxetine, calcium and placebo groups, 8, 11 and 12 participants remained in the trial until Visit 5.
Measure: Number; unit: proportion of participants
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 8 | 11 | 12
proportion of participants | 0.75 | 0.36 | 0.17
Statistical Analysis 1: Comparison: I: Fluoxetine vs II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.04, Chi-squared

7. Primary Outcome: Comparison of the Change in IDS Symptom Scores Among Groups
Description: IDS = Inventory of Depressive Symptomatology: measures depressive symptoms during the previous premenstrual phase with high internal consistency: sum of responses to 28 of 30 possible items each scored 0 to 3 points with total scoring (0=no symptoms, 84=most severe). This outcome is a measure of effect size between the two trial groups and the placebo group, with the placebo effect size value used as a reference.
Time Frame: over duration of treatment, 4 menstrual cycles averaging 4 months after baseline visit
Population: Intention to treat cohort.
Measure: Mean (Standard Deviation); unit: units on IDS scale
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 13 | 13 | 13
units on IDS scale
  Visit 1 | 31.85 (9.14) | 30.92 (7.62) | 28.85 (9.97)
  Visit 2 | 14.08 (9.53) | 25.77 (7.74) | 20.69 (12.20)
  Visit 3 | 11.44 (7.94) | 18.55 (10.40) | 20.15 (14.25)
  Visit 4 | 11.78 (8.50) | 18.50 (9.01) | 16.46 (11.00)
  Visit 5 | 10.00 (6.41) | 19.55 (9.04) | 18.08 (9.17)
Statistical Analysis 1: Comparison: I: Fluoxetine vs III: Placebo; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis; Slope = -2.63, 95% CI 2-sided [-5.51 to 0.24] — Slope represents average change in fluoxetine group IDS score as compared to placebo
Statistical Analysis 2: Comparison: II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis; Slope = -0.10, 95% CI 2-sided [-2.85 to 2.65] — Slope represents average change in calcium group IDS scores as compared to placebo
Statistical Analysis 3: Comparison: I: Fluoxetine vs III: Placebo; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis; Cohen's d effect size = 1.15 — Cohen's d effect sizes were calculated by subtracting the difference between changes in the fluoxetine group between visits 1 and 5 and changes in the placebo group between Visits 1 and 5, divided by the std dev in the placebo group at Visit 5
Statistical Analysis 4: Comparison: II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis; Cohen's d effect size = 0.10 — Cohen's d effect sizes were calculated by subtracting the difference between changes in the calcium group between visits 1 and 5 and changes in the placebo group between Visits 1 and 5, divided by the std dev in the placebo group at Visit 5

8. Primary Outcome: Comparison of the Change in PMTS Symptom Scores Among Groups
Description: PMTS = Premenstrual Tension Syndrome (Observer Rating) Scale: a clinician-administered retrospective scale developed for the study of PMS, a sum of responses to 10 items each with 4 points (0=no symptoms, 40=most severe). This outcome is a measure of effect size between the two trial groups and the placebo group, with the placebo effect size value used as a reference.
Time Frame: over duration of treatment, 4 menstrual cycles averaging 4 months after baseline visit
Population: Intention to treat cohort.
Measure: Mean (Standard Deviation); unit: units on PMTS scale
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 13 | 13 | 13
units on PMTS scale
  Visit 1 | 24.15 (5.40) | 21.58 (3.73) | 20.85 (6.62)
  Visit 2 | 11.15 (5.77) | 18.54 (5.36) | 16.00 (8.15)
  Visit 3 | 10.33 (6.40) | 13.36 (5.75) | 16.38 (10.52)
  Visit 4 | 12.11 (7.13) | 12.83 (4.73) | 12.77 (8.21)
  Visit 5 | 10.13 (3.56) | 11.91 (4.48) | 14.58 (7.58)
Statistical Analysis 1: Comparison: I: Fluoxetine vs III: Placebo; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis; Slope = -1.63, 95% CI 2-sided [-3.60 to 0.34] — Slope represents average change in fluoxetine group PMTS scores as compared to placebo
Statistical Analysis 2: Comparison: II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.40, Mixed Models Analysis; Slope = -0.81, 95% CI 2-sided [-2.71 to 1.09] — Slope represents average change in calcium group PMTS scores as compared to placebo
Statistical Analysis 3: Comparison: I: Fluoxetine vs III: Placebo; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis; Cohen's d effect size = 1.06 — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 4: Comparison: II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.40, Mixed Models Analysis; Cohen's d effect size = 0.37 — [estimate comment as in outcome 7, analysis 4]

9. Primary Outcome: Comparison of the Change in CGI-S Symptom Scores Among Groups
Description: CGI-S = Clinical Global Impression-Severity: a severity scale widely used in psychopharmacology research (1=normal not at all ill, 7=among most extremely ill). This outcome is a measure of effect size between the two trial groups and the placebo group, with the placebo effect size value used as a reference.
Time Frame: over duration of treatment, 4 menstrual cycles averaging 4 months after baseline visit
Population: Intention to treat cohort.
Measure: Mean (Standard Deviation); unit: units on CGI-S scale
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 13 | 13 | 13
units on CGI-S scale
  Visit 1 | 4.92 (0.95) | 4.46 (1.27) | 4.15 (1.28)
  Visit 2 | 2.54 (1.13) | 4.23 (1.01) | 3.38 (1.66)
  Visit 3 | 2.33 (1.00) | 3.00 (1.10) | 3.38 (1.98)
  Visit 4 | 2.56 (1.13) | 2.73 (0.90) | 2.92 (1.50)
  Visit 5 | 2.50 (0.76) | 2.91 (1.04) | 3.17 (1.47)
Statistical Analysis 1: Comparison: I: Fluoxetine vs III: Placebo; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis; Slope = -0.35, 95% CI 2-sided [-0.73 to 0.03] — Slope represents average change in fluoxetine group CGI-S scores as compared to placebo
Statistical Analysis 2: Comparison: II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.36, Mixed Models Analysis; Slope = -0.17, 95% CI 2-sided [-0.54 to 0.20] — Slope represents average change in calcium group CGI-S scores as compared to placebo
Statistical Analysis 3: Comparison: I: Fluoxetine vs III: Placebo; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis; Cohen's d effect size = 0.92 — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 4: Comparison: II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.36, Mixed Models Analysis; Cohen's d effect size = 0.44 — [estimate comment as in outcome 7, analysis 4]

10. Primary Outcome: Comparison of the Change in DRSP Symptom Scores Among Groups
Description: DRSP = Daily Record of Severity of Problems, which combines responses to 21 items each with scale: 1=no symptoms, 6=extreme. This outcome is a measure of effect size between the two trial groups and the placebo group, with the placebo effect size value used as a reference.
Time Frame: over duration of treatment, 4 menstrual cycles averaging 4 months after baseline visit
Population: Intention to treat cohort.
Measure: Mean (Standard Deviation); unit: units on DRSP scale
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 13 | 13 | 13
units on DRSP scale
  Visit 1 | 2.16 (0.86) | 1.12 (0.38) | 1.29 (0.60)
  Visit 2 | 0.97 (0.72) | 0.76 (0.78) | 0.93 (0.54)
  Visit 3 | 0.27 (0.78) | 0.61 (0.78) | 1.19 (1.06)
  Visit 4 | 0.72 (0.78) | 0.51 (0.33) | 0.59 (0.63)
  Visit 5 | 0.44 (0.34) | 0.75 (0.42) | 0.74 (0.54)
Statistical Analysis 1: Comparison: I: Fluoxetine vs III: Placebo; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Slope = -0.28, 95% CI 2-sided [-0.53 to -0.04] — Slope represents average change in fluoxetine group DRSP scores as compared to placebo
Statistical Analysis 2: Comparison: II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.58, Mixed Models Analysis; Slope = 0.06, 95% CI 2-sided [-0.16 to 0.28] — Slope represents average change in calcium group DRSP scores as compared to placebo
Statistical Analysis 3: Comparison: I: Fluoxetine vs III: Placebo; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Cohen's d effect size = 2.08 — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 4: Comparison: II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.58, Mixed Models Analysis; Cohen's d effect size = 0.18 — [estimate comment as in outcome 7, analysis 4]

11. Primary Outcome: Comparison of the Change in CGI Improvement Scores Among Groups
Description: CGI-I = Clinical Global Impression Improvement: the improvement subscale of CGI measuring change at each visit as compared to visit 1 (1=very much improved, 7=very much worse). This outcome is a measure of effect size between the two trial groups and the placebo group, with the placebo effect size value used as a reference.
Time Frame: over duration of treatment, 4 menstrual cycles averaging 4 months after baseline visit
Population: Intention to treat cohort.
Measure: Mean (Standard Deviation); unit: units on CGI Improvement scale
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Number analyzed (Participants) | 13 | 13 | 13
units on CGI Improvement scale
  Visit 1 | NA (NA) — at first visit, improvement since last visit cannot be scored | NA (NA) — at first visit, improvement since last visit cannot be scored | NA (NA) — at first visit, improvement since last visit cannot be scored
  Visit 2 | 2.23 (0.83) | 3.46 (0.78) | 3.00 (1.35)
  Visit 3 | 1.67 (0.87) | 2.30 (0.82) | 3.08 (1.50)
  Visit 4 | 1.75 (1.16) | 2.36 (1.03) | 2.77 (1.17)
  Visit 5 | 1.88 (0.64) | 2.45 (0.82) | 2.83 (1.19)
Statistical Analysis 1: Comparison: I: Fluoxetine vs III: Placebo; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Slope = -1.03, 95% CI 2-sided [-1.70 to -0.35] — Slope represents average change in fluoxetine group CGI Improvement scores as compared to placebo
Statistical Analysis 2: Comparison: II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.54, Mixed Models Analysis; Slope = -0.20, 95% CI 2-sided [-0.86 to 0.46] — Slope represents average change in calcium group CGI Improvement scores as compared to placebo
Statistical Analysis 3: Comparison: I: Fluoxetine vs III: Placebo; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Cohen's d effect size = 0.80 — Cohen's d effect sizes were calculated by subtracting the difference between changes in the fluoxetine group between visits 2 and 5 and changes in the placebo group between Visits 2 and 5, divided by the std dev in the placebo group at Visit 5
Statistical Analysis 4: Comparison: II: Calcium vs III: Placebo; Test type: Superiority or Other; p = 0.54, Mixed Models Analysis; Cohen's d effect size = 0.32 — Cohen's d effect sizes were calculated by subtracting the difference between changes in the calcium group between visits 2 and 5 and changes in the placebo group between Visits 2 and 5, divided by the std dev in the placebo group at Visit 5

ADVERSE EVENTS:
Time Frame: From patient randomization to completion of study
Description: Final adverse event data were only available for the 32 patients randomized at the Yale site. There were no severe adverse events by self-report. Events were uncommon and occurred in all 3 groups with a numerically higher number in the calcium group.
Arm/Group | I: Fluoxetine | II: Calcium | III: Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 4/10 | 8/11 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I: Fluoxetine (N=10) | II: Calcium (N=11) | III: Placebo (N=11)
Feeling spacy (General disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal ache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Burping (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Difficulty Concentrating (General disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cramps (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased sex drive (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (General disorders) | 1 (1) | 2 (2) | 0 (0)
Dry mouth (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 3 (3) | 2 (2)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Sweating (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (General disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No